CLINICAL TRIAL: NCT04586517
Title: Effects of Heavy-load Resistance Training During (Neo-)Adjuvant Chemotherapy on Muscle Cellular Outcomes in Women With Breast Cancer
Brief Title: Effect of Heavy-load Resistance Training During Chemotherapy on Muscle Cellular Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Collaborators: Swedish Cancer Society (Other); Norwegian Cancer Society (Other); Norwegian School of Sport Sciences (Other); University of Agder (Other); Rigshospitalet, Denmark (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Karin Nordin, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01097
Record Dates: First submitted 2020-09-25; First posted 2020-10-14 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer Female
Keywords: Breast cancer; Resistance training; Chemotherapy; Randomized controlled trial; Muscle biopsies; Cross-sectional fiber area
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise; Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive supervised heavy-load resistance training twice a week during treatment with chemotherapy (approximately 16-weeks). After end of chemotherapy, participants will be encouraged to continue the training program and are provided with 12-month membership at a local gym.
  Interventions: Other: Heavy-load resistance training
- Control group (Active Comparator): Participants will be encouraged to continue with their usual activities during chemotherapy and not start resistance training (approximately 16-weeks). After end of chemotherapy participants will be offered to attend a 2-week introduction to the strength-training program and provided with a 12-month membership at a local gym.
  Interventions: Other: Control

INTERVENTIONS:
Other: Heavy-load resistance training — Supervised heavy-load resistance training during chemotherapy treatment
  Other Names: Physical exercise; Physical training
  Arms: Intervention group
Other: Control — Activity as usual during chemotherapy
  Other Names: usual care
  Arms: Control group

SUMMARY:
(Neo-)adjuvant chemotherapy for breast cancer is known to have a negative impact on muscle tissue resulting in reduced aerobic fitness, skeletal muscle mass and strength. Physical exercise during treatment may counteract some of these negative effects. However, the effects of resistance training alone have never been explored. The present study aims to investigate if heavy-load resistance training during (neo-)adjuvant chemotherapy counteracts negative effects on skeletal muscle in women diagnosed with breast cancer. The hypothesis is that (neo-)adjuvant treatment with chemotherapy will reduce muscle fiber size, impair mitochondrial function and increase indicators of cellular stress and that resistance training during treatment will counteract these negative effects. Fifty women recently diagnosed with breast cancer scheduled to start (neo-)adjuvant chemotherapy will be randomized to either an intervention group or a control group. The intervention group will perform supervised heavy-load resistance training twice a week over the course of chemotherapy (approximately 16-weeks) whereas the control group will be encouraged to continue with their usual activities. To increase interest in participation, controls will be invited to a 2-week introduction to the same resistance-training program as the intervention group following completion of chemotherapy. Muscle biopsies from m. vastus lateralis will be collected before the first cycle of chemotherapy, after chemotherapy, and 6 months later (6-month follow-up) for assessment of muscle cellular outcomes. Results from this intervention will provide further knowledge on how chemotherapy affects muscle tissue and how resistance training may counteract immediate and long-term treatment side effects. Results from this intervention will also contribute with knowledge about how to improve exercise programs that are effective for women undergoing chemotherapy against breast cancer.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of heavy-load resistance training on muscle cellular outcomes in women with breast cancer undergoing (neo-)adjuvant chemotherapy.

More specifically, the investigators' objectives are to

1. Investigate the effects of a heavy-load resistance training intervention on skeletal muscle fiber cross-sectional area.
2. Investigate the effects of a heavy-load resistance training intervention on regulators of muscle fiber size, muscle fiber function, cellular stress and mitochondrial function.
3. Investigate the effects of chemotherapy on skeletal muscle fiber cross-sectional area, regulators of muscle fiber size, muscle fiber function, cellular stress and mitochondrial function.
4. Explore the effects of heavy-load resistance training on the expression levels of myokines.

This study is a two-armed randomized controlled trial with follow-up at six months. With this design, the investigators can study the main effect and interactions between factors (groups). Participants will be randomized to either an intervention group or a control group.

Participants recently diagnosed with breast cancer will be recruited from Uppsala University Hospital. Based on power calculations, 50 participants will be included. Data will be collected before the first cycle of chemotherapy, after chemotherapy, and 6 months later (6-month follow-up.

Participants in the intervention group will perform supervised heavy-load resistance training twice a week from the week following the start of chemotherapy and throughout the course of treatment, approximately 16 weeks. Sessions will be performed at a public gym and led by trained coaches. The following six exercises will be included in the program: seated leg-press, seated chest press, seated leg-curl, seated row and seated leg-extension performed in machines and seated overhead-press using dumbbells. The first two weeks of the program represent familiarization to the training protocol and 1 RM (Repetition Maximum) tests. During this period, the participants will perform exercises at a light load. After the first 1 RM-test, training will progress in sets and training load before testing of 6- and 10 RM which will provide the participants with individualized loads. Rest periods between sets will be two (6 RM training load) and one minute (10 RM training load) for the two different sessions, respectively. The training load will be adjusted throughout the intervention period. Participants in the control group are encouraged to continue with their activity as usual i.e. maintain their habitual physical activity level and not initiate resistance training during chemotherapy. To increase interest in participation, controls will be invited to a 2-week introduction to the same resistance-training program as the intervention group following completion of chemotherapy and offered a 12-month membership at a local gym, free of charge.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with stage I-III breast cancer
* literate in Swedish
* scheduled to undergo (neo-)adjuvant chemotherapy with a combination of taxanes and anthracyclines or only one of these treatments

Exclusion Criteria:

* unable to perform basic activities of daily living
* cognitive disorders or severe emotional instability
* other disabling comorbidities that might hamper physical training (e.g. severe heart failure, chronic obstructive pulmonary disease, orthopedic conditions, and neurological disorders)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in muscle fiber cross-sectional area | From baseline to the 16 week time-point
  Change from baseline in muscle fiber cross-sectional area at 16 weeks. Through immunohistochemical staining of muscle fiber cross-sections will muscle fiber area be assessed for type 1 and type 2 muscle fibers

SECONDARY OUTCOMES:
Assessment of changes in muscle fiber cross-sectional area | From baseline to 6-month follow-up
  Change from baseline in muscle fiber cross-sectional area at 6-month follow-up. Through immunohistochemical staining of muscle fiber cross-sections will muscle fiber area be assessed for type 1 and type 2 muscle fibers
Assessment of changes in satellite cell content in muscle fiber cross-sections | From baseline to the 16 week time-point and from baseline to 6-month follow-up
  Change from baseline in satellite cell content in muscle fiber cross-sections at 16 weeks and at 6-month follow-up. Through immunohistochemical staining of muscle fiber cross-sections will satellite cell content be assessed per muscle fiber
Assessment of changes in myonuclei content in muscle fiber cross-sections | From baseline to the 16 week time-point and from baseline to 6-month follow-up
  Change from baseline in myonuclei content in muscle fiber cross-sections at 16 weeks and at 6-month follow-up. Through immunohistochemical staining of muscle fiber cross-sections will myonuclei content be assessed per muscle fiber
Assessment of protein levels of regulators of muscle fiber size (proteins involved in muscle protein synthesis and protein degradation (e.i. mTOR, MuRF, S6K1, p70S6k) | From baseline to the 16 week time-point and from baseline to 6-month follow-up
  Change from baseline in protein levels of regulators of muscle fiber size at 16 weeks and at 6-month follow-up. Proteins involved in regulation of muscle size (muscle protein synthesis and protein degradation) will be assessed in muscle homogenate using Western blot analysis
Assessment of changes in protein levels of regulators of muscle fiber cellular stress (Heat Shock proteins: Hsp 27, αB-crystalline, Hsp 60 and Hsp 70) | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in protein levels of regulators of muscle fiber cellular stress at 16 weeks and at 6-month follow-up. Proteins involved in protection against cellular stress will be assessed in muscle homogenate using Western blot analysis
Assessment of changes in protein levels of regulators of mitochondrial function (Citric syntase, Cox 4 and HAD) | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in protein levels of regulators of muscle fiber mitochondrial function at 16 weeks and at 6-month follow-up. Proteins involved in protection/enzymes involved in mitochondrial function will be assessed in muscle homogenate using Western blot analysis
Assessment of changes in myokines with potential anti-tumor effects | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in protein levels of myokines with potential anti-tumor effects at 16 weeks and at 6-month follow-up. Myokines assossiated with potential anti-tumor effects will be assessed in muscle homogenate using Western blot analysis
Changes in muscle strength | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Maximal upper- and lower extremity muscle strength will be assessed as one repetition maximum in seated chest-press and seated single-leg press
Cardiorespiratory fitness | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Cardiorespiratory fitness will be assessed as maximal oxygen uptake during maximal walking/running until exhaustion on a treadmill

OTHER OUTCOMES:
Assessment of changes fat free mass | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in fat free mass at 16 weeks and at 6-month follow-up will be assessed using air displacement plethysmography and bioelectrical impedance analysis.
Assessment of changes in fat mass | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in fat mass at 16 weeks and at 6-month follow-up will be assessed using air displacement plethysmography and bioelectrical impedance analysis. From this analysis fat free mass, fat mass, body density and body water content will be derived
Assessment of blood lipids | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in blood lipids at 16 weeks and at 6-month follow-up, assessed in blood serum and plasma using ELISA methods.
Assessment of C-reactive protein | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in C-reactive protein at 16 weeks and at 6-month follow-up, assessed in blood serum and plasma using ELISA methods.
Assessment of creatine kinase-myocardial band | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in creatine kinase-myocardial band at 16 weeks and at 6-month follow-up, assessed in blood serum and plasma using ELISA methods.
Assessment of blood glucose | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in blood glucose at 16 weeks and at 6-month follow-up, assessed in blood serum and plasma using ELISA methods.
Assessment of serum cortisol | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in serum cortisol at 16 weeks and at 6-month follow-up, assessed in blood serum and plasma using ELISA methods.
Assessment of hemoglobin | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in hemoglobin at 16 weeks and at 6-month follow-up, assessed in blood serum and plasma using ELISA methods.
Assessment of changes in quality of life | From baseline to the 16 week time-point and from baseline to the 6-month follow-up
  Change from baseline in quality of life at 16 weeks and at 6-month follow-up using The European Organization for Research and Treatment of Cancer (EORTC)EORTC-QLQ30
Assessment of changes in fatigue | From baseline to the 16 week time point and from baseline to the 6-month follow-up
  Change from baseline in fatigue at 16 weeks and at 6-month follow-up using Multi Dimensional Fatigue Inventory (MFI)
Assessment of physical activity, defined as minutes spent in moderate-to-vigorous intensity activity | Measurement at three time points, baseline, 16 weeks and 6-month follow-up
  Assessment of physical activity, assessed by the SenseWear Armband activity monitoring device. The purpose is to monitor and to be able to adjust for the participants' physical activity outside the intervention as a possible confounder. A SenseWear Armband is worn for 7 consecutive days at three time points (baseline, 16 weeks and 6-month follow-up).
Adverse events | Through study completion, an average of 1 year
  Adverse events from training session and muscle biopsy sampling will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Truls Raastad, PhD, Principal Investigator — Norweigan School of Sport Sciences; Karin Nordin, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Mazzoni AS, Strandberg E, Borjeson S, Sjovall K, Berntsen S, Demmelmaier I, Nordin K. Reallocating sedentary time to physical activity: effects on fatigue and quality of life in patients with breast cancer in the Phys-Can project. Support Care Cancer. 2023 Feb 4;31(2):151. doi: 10.1007/s00520-023-07614-9. PMID 36738358
- [Derived] Strandberg E, Vassbakk-Svindland K, Henriksson A, Johansson B, Vikmoen O, Kudren D, Schauer T, Lindman H, Warnberg F, Berntsen S, Demmelmaier I, Nordin K, Raastad T. Effects of heavy-load resistance training during (neo-)adjuvant chemotherapy on muscle cellular outcomes in women with breast cancer. Medicine (Baltimore). 2021 Mar 12;100(10):e24960. doi: 10.1097/MD.0000000000024960. PMID 33725859